CLINICAL TRIAL: NCT02618915
Title: Phase I/II Open-Label Safety and Dose Finding Study of Adeno-Associated Virus (AAV) rh10-Mediated Gene Transfer of Human Factor IX in Adults With Moderate/Severe to Severe Hemophilia B
Brief Title: Safety and Dose Finding Study of DTX101 (AAVrh10FIX) in Adults With Moderate/Severe to Severe Hemophilia B
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision; not due to any safety concerns related to DTX101.
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101HEMB01
Record Dates: First submitted 2015-11-23; First posted 2015-12-02 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Hemophilia B
Keywords: gene therapy; Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DTX101, Cohort 1 (Experimental): a single peripheral intravenous (IV) infusion of 1.6 x 10^12 genome copies (GC)/kg DTX101
  Interventions: Genetic: DTX101
- DTX101, Cohort 2 (Experimental): a single peripheral IV infusion of 5.0 x 10^12 GC/kg DTX101
  Interventions: Genetic: DTX101

INTERVENTIONS:
Genetic: DTX101 — solution for IV infusion
  Other Names: non-replicating recombinant AAVrh10 encoding human FIX (hFIX); AAVrh10FIX

SUMMARY:
A Phase 1/2, open-label, dose-finding safety study of single ascending doses of DTX101 in adult males with moderate/severe to severe hemophilia B.

DETAILED DESCRIPTION:
Hemophilia B is an X-linked recessive genetic bleeding disorder caused by mutations in the factor IX (FIX) gene. FIX is produced in the liver and is critical for fibrin clot formation. Hemophilia B is characterized by frequent, spontaneous internal bleeding that can lead to chronic arthropathy (joint damage), intracranial hemorrhage, and even death. In patients with moderate/severe to severe hemophilia B, the majority of bleeding episodes occur in the joints and, if not treated, lead to debilitating damage and a decreased quality of life.

This study will evaluate the safety and efficacy of the adeno-associated virus (AAV) to deliver human factor IX (hFIX) gene, the healthy gene necessary to make FIX, to the liver where FIX is normally produced. This study will determine if AAVrh10 can produce clinically meaningful FIX levels in patients with moderately/severe or severe hemophilia B.

This study was previously posted by Dimension Therapeutics, which has been acquired by Ultragenyx in November 2017.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥ 18 years of age.
2. Moderate/severe or severe hemophilia B (baseline FIX activity ≤ 2% of normal or documented history of FIX activity ≤2%).
3. At least 3 bleeding episodes per year that require on-demand treatment with FIX OR are treated with a prophylactic regimen of FIX.
4. At least 100 days exposure history to FIX.
5. No documented history of inhibitors (neutralizing antibodies) to exogenous FIX.
6. No known allergic reaction to exogenous FIX or any component of DTX101.
7. Willing to stop prophylactic treatment with recombinant FIX at specified time points during the study.

Exclusion Criteria:

1. History of significant liver disease (ie, portal hypertension).
2. Significant hepatic inflammation or cirrhosis.
3. Evidence of active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
4. History of human immunodeficiency virus (HIV) infection AND any of the following: CD4+ cell count < 350 cells/mm^3, change in antiretroviral therapy regimen within 6 months prior to Day 0, or plasma viral load > 200 copies/mL, on 2 separate occasions, as measured by polymerase chain reaction.
5. Anti-AAVrh10 neutralizing antibody titer > 1:5.
6. Participation (current or previous) in another gene therapy study.
7. Participation in another investigational medicine study within 3 months before screening.

NOTE: Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (9):
- United States (6):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Orthopaedic Institute for Children, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Hospital and Health Systems, Michigan Clinical Research Unit, Ann Arbor, Michigan
  - Vanderbilt Hemostasis-Thrombosis Clinic, Nashville, Tennessee
- Specialized Hospital for Active Treatment for Hematological Disease, Sofia, Bulgaria
- United Kingdom (2):
  - Basingstoke and North Hampshire Hospital, Haemophilia, Haemostasis and Thrombosis Centre, Basingstoke, Hampshire
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Pipe S, Poma A, Rajasekhar A, Everington T, Sankoh S, Allen J, Cataldo J, Crombez E. Gene therapy for hemophilia B: results from the phase 1/2 101HEMB01/02 studies. Blood Adv. 2025 Jun 24;9(12):2980-2987. doi: 10.1182/bloodadvances.2024015184. PMID 40197980

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DTX101, Cohort 1 | DTX101, Cohort 2
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DTX101, Cohort 1: a single peripheral IV infusion of 1.6 x 10^12 GC/kg DTX101
- Total: Total of all reporting groups
Arm/Group | DTX101, Cohort 1 | DTX101, Cohort 2 | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Customized [Number; unit: participants]
  18-49 years | 0 | 3 | 3
  50-84 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Factor IX (FIX) Activity [Mean (Standard Deviation); unit: IU/dL] — The documented history or measurement before the Day 0 visit following the appropriate washout was used for the baseline values of FIX activity.
  IU/dL | 1.67 (0.577) | 0.87 (0.709) | 1.27 (0.566)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Treatment-Related Adverse Events (TEAEs), and Serious AEs (SAEs)
Description: An AE was defined as any untoward medical occurrence in a participant enrolled into this study (from the time the participant signed the informed consent form until his or her exit from the study), regardless of its causal relationship to study treatment. A TEAE was defined as any event not present before exposure to study product or any event already present that worsened in severity or increased in frequency after exposure to study product.
Time Frame: up to 52 weeks after dosing (Cohort 1) or 44 weeks after dosing (Cohort 2)
Population: Safety Set: all participants who received DTX101 including participants who received a partial dose or failed infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | DTX101, Cohort 1 | DTX101, Cohort 2
Number analyzed (Participants) | 3 | 3
Participants
  All TEAEs | 3 | 3
  All Serious TEAEs | 1 | 0

2. Primary Outcome: Change From Baseline in FIX Activity at Week 6
Description: Peak plasma level of FIX after IV administration as determined by the activated partial thromboplastin time (aPTT) clot-based assay. Change from baseline: postbaseline value - baseline value. For the change from baseline, only participants with a value at both baseline visit and the specific postbaseline visit were included.
Time Frame: Baseline, Week 6
Population: As Treated Set: all participants who received any amount of DTX101.
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | DTX101, Cohort 1 | DTX101, Cohort 2
Number analyzed (Participants) | 3 | 3
IU/dL | 5.00 (1.732) | 9.80 (4.687)

3. Secondary Outcome: Annualized Bleeding Rate
Description: The number of bleeding episodes per participant was recorded, and the annualized number of bleeding episodes was calculated.
Time Frame: Week 0 to Week 52
Population: As Treated Set: all participants who received any amount of DTX101.
Measure: Mean (Standard Deviation); unit: bleeding episodes/year
Groups:
- DTX101, Dose 1: 1.6 x 10^12 genome copies (GC)/kg DTX101
- DTX101, Dose 3: 5.0 x 10^12 GC/kg DTX101
Arm/Group | DTX101, Dose 1 | DTX101, Dose 3
Number analyzed (Participants) | 3 | 3
bleeding episodes/year | 8.7 (5.53) | 5.0 (1.00)

4. Secondary Outcome: Change From Baseline in FIX Activity Over Time
Description: Peak plasma level of FIX after IV administration as determined by the aPTT clot-based assay. Change from baseline: postbaseline value - baseline value. For the change from baseline, only participants with a value at both baseline visit and the specific postbaseline visit were included. Participants were not required to stop prophylactic treatment with recombinant FIX until after Week 4 and may have been restarted on their prophylactic recombinant FIX treatment after Week 14.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 12, 16, 24, 32, 40, End of Study (Week 52 for Cohort 1, Week 44 for Cohort 2)/Early Withdrawal
Population: As Treated Set: all participants who received any amount of DTX101.
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | DTX101, Cohort 1 | DTX101, Cohort 2
Number analyzed (Participants) | 3 | 3
IU/dL
  Week 2 | 16.33 (14.503) | 10.13 (7.988)
  Week 4 | 8.67 (7.234) | 14.47 (10.835)
  Week 6 | 5.00 (1.732) | 9.80 (4.687)
  Week 8 | 14.67 (17.786) | 11.80 (6.646)
  Week 12 | 11.33 (4.933) | 5.80 (2.207)
  Week 16 | 7.67 (3.215) | 5.47 (3.066)
  Week 24 | 2.33 (1.528) | 2.47 (2.214)
  Week 32 | 9.33 (11.846) | 10.13 (2.702)
  Week 40 | 15.33 (23.965) | 12.80 (16.008)
  End of Study/Early Withdrawal | 1.67 (0.577) | 22.47 (1.380)

5. Secondary Outcome: Annualized FIX Replacement Therapy
Description: The use of on-demand FIX replacement therapy was recorded by dose (IU/kg) administered, and the annualized use of FIX replacement therapy was calculated. Participants were not required to stop prophylactic treatment with recombinant FIX until after Week 4 and may have been restarted on their prophylactic recombinant FIX treatment after Week 14.
Time Frame: Week 0 to Week 52
Population: As Treated Set: all participants who received any amount of DTX101.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | DTX101, Cohort 1 | DTX101, Cohort 2
Number analyzed (Participants) | 3 | 3
IU/kg | 350115.2 (522106.19) | 64246.5 (805.34)

6. Secondary Outcome: Number of Participants With Neutralizing Antibodies to FIX (FIX Inhibitors)
Description: The development of neutralizing antibodies to FIX (FIX inhibitors), as determined by a Bethesda assay. A value of < 0.3 inhibitor units was considered to be no neutralizing antibodies.
Time Frame: Day 0 (predose), Weeks 6, 8, 16, 32, 40, End of Study (Week 52 for Cohort 1, Week 44 for Cohort 2)/Early Withdrawal
Population: As Treated Set: all participants who received any amount of DTX101.
Measure: Count of Participants; unit: Participants
Arm/Group | DTX101, Cohort 1 | DTX101, Cohort 2
Number analyzed (Participants) | 3 | 3
Participants
  Day 0 (predose) | 0 | 0
  Week 6 | 0 | 0
  Week 8 | 0 | 0
  Week 16 | 0 | 0
  Week 32 | 0 | 0
  Week 40 | 0 | 0
  End of Study/Early Withdrawal | 0 | 0

7. Secondary Outcome: Number of Participants With Cell-Mediated Immune Response to FIX
Description: The development of a cell-mediated immune response to FIX, as determined by enzyme-linked immunospot assay (ELISPOT).
Time Frame: Day 0 (predose), Weeks 6, 8, 12, 16, 32, 40, 48, End of Study (Week 52 for Cohort 1, Week 44 for Cohort 2)/Early Withdrawal
Population: Safety Set: all participants who received DTX101 including subjects who received a partial dose or failed infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | DTX101, Cohort 1 | DTX101, Cohort 2
Number analyzed (Participants) | 3 | 3
Participants
  Day 0 (predose) | 0 | 0
  Week 6 | 0 | 0
  Week 8 | 0 | 0
  Week 12 | 0 | 0
  Week 16 | 0 | 0
  Week 32 | 0 | 0
  Week 40 | 0 | 0
  Week 48 | 0 | 0
  End of Study/Early Withdrawal | 0 | 0

8. Secondary Outcome: Number of Participants Responding to the EuroQoL-5D-5 Level (EQ-5D-5L) Questionnaire
Description: EQ-5D-5L is a standardized, subject-rated instrument for use as a measure of health outcomes. The EQ 5D-5L includes 2 components: the EQ-5D-5L descriptive system and the EQ visual analogue scale (EQ-VAS). The EQ-5D-5L descriptive system provides a profile of the participant's health state in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each dimension, the participant is instructed to indicate whether he or she has "no problems" (1), "some problems" (2), or "severe problems" (3).
Time Frame: Baseline (Day 0 predose), Weeks 24, 36, 48, End of Study/Early Withdrawal (up to Week 52)
Population: Safety Set: all participants who received DTX101 including participants who received a partial dose or failed infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | DTX101, Cohort 1 | DTX101, Cohort 2
Number analyzed (Participants) | 3 | 3
Participants
  Day 0 | 3 | 3
  Week 24 | 3 | 3
  Week 36 | 3 | 2
  Week 48 | 2 | 1
  End of Study/Early Withdrawal | 2 | 0

9. Secondary Outcome: Number of Participants Responding to the Haemophilia-Specific Quality of Life Questionnaire
Description: The Haemophilia-Specific Quality of Life questionnaire asks subjects about their perceptions of their health and treatment. The questionnaire is divided into the following 10 dimensions: physical health, feelings, view of themselves, sports & leisure, work & school, dealing with hemophilia, treatment, future, family planning, and partnership & sexuality. Questions are based on a 5-point Likert-scale (1=never, 2=rarely, 3=sometimes, 4=often, 5=all the time). If the question does not apply to the subject, the "not applicable" response is allowed in 3 of the domains (sport & leisure, work & school, family planning). Positively worded items need to be re-coded and domains will be transformed ranging from 0 to 100; higher domain and total scores indicating a higher impairment of health-related quality of life.
Time Frame: Baseline (Day 0 predose), Weeks 24, 36, 48, End of Study/Early Withdrawal (up to Week 52)
Population: Safety Set: all participants who received DTX101 including participants who received a partial dose or failed infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | DTX101, Cohort 1 | DTX101, Cohort 2
Number analyzed (Participants) | 3 | 3
Participants
  Day 0 | 3 | 3
  Week 24 | 3 | 3
  Week 36 | 3 | 2
  Week 48 | 2 | 1
  End of Study/Early Withdrawal | 2 | 0

10. Secondary Outcome: Average Weekly Use of FIX Replacement Therapy
Description: The use of on-demand FIX replacement therapy was recorded by dose (IU/kg) administered and the average weekly use of FIX replacement therapy was calculated. Participants were not required to stop prophylactic treatment with recombinant FIX until after Week 4 and may have been restarted on their prophylactic recombinant FIX treatment after Week 14.
Time Frame: Baseline (Screening), Week 0 through Week 52
Population: As Treated Set: all participants who received any amount of DTX101, with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | DTX101, Cohort 1 | DTX101, Cohort 2
Number analyzed (Participants) | 3 | 3
IU/kg
  Baseline | 9659.1 (12502.19) | 5037.2 (3502.95)
  Week 0 to 2: number analyzed (Participants) | 2 | 1
  Week 0 to 2 | 12120.0 (11144.00) | 5000.0 (NA) — Only 1 participant analyzed at this time point.
  Week 3 to 4: number analyzed (Participants) | 1 | 1
  Week 3 to 4 | 24000.0 (NA) — Only 1 participant analyzed at this time point. | 7000.0 (NA) — Only 1 participant analyzed at this time point.
  Week 5 to 6: number analyzed (Participants) | 2 | 1
  Week 5 to 6 | 9068.5 (10611.55) | 3000.0 (NA) — Only 1 participant analyzed at this time point.
  Week 7 to 8: number analyzed (Participants) | 2 | 0
  Week 7 to 8 | 5120.0 (1244.51) |
  Week 9 to 10: number analyzed (Participants) | 1 | 0
  Week 9 to 10 | 32000.0 (NA) — Only 1 participant analyzed at this time point. |
  Week 11 to 12: number analyzed (Participants) | 3 | 0
  Week 11 to 12 | 8076.7 (10325.91) |
  Week 13 to 14: number analyzed (Participants) | 1 | 0
  Week 13 to 14 | 12000.0 (NA) — Only 1 participant analyzed at this time point. |
  Week 15 to 16: number analyzed (Participants) | 1 | 0
  Week 15 to 16 | 16000.0 (NA) — Only 1 participant analyzed at this time point. |
  Week 17 to 18: number analyzed (Participants) | 1 | 2
  Week 17 to 18 | 8000.0 (NA) — Only 1 participant analyzed at this time point. | 3375.0 (883.88)
  Week 19 to 20: number analyzed (Participants) | 1 | 1
  Week 19 to 20 | 12000.0 (NA) — Only 1 participant analyzed at this time point. | 8000.0 (NA) — Only 1 participant analyzed at this time point.
  Week 21 to 22: number analyzed (Participants) | 3 | 0
  Week 21 to 22 | 7832.8 (3057.68) |
  Week 23 to 24: number analyzed (Participants) | 2 | 0
  Week 23 to 24 | 8782.5 (10207.09) |
  Week 25 to 26: number analyzed (Participants) | 2 | 2
  Week 25 to 26 | 8902.5 (4380.53) | 5445.0 (3952.73)
  Week 27 to 28: number analyzed (Participants) | 2 | 2
  Week 27 to 28 | 8120.0 (5487.15) | 4725.0 (1025.30)
  Week 29 to 30: number analyzed (Participants) | 2 | 2
  Week 29 to 30 | 12120.0 (11144.00) | 2250.0 (353.55)
  Week 31 to 32: number analyzed (Participants) | 1 | 2
  Week 31 to 32 | 28000.0 (NA) — Only 1 participant analyzed at this time point. | 2750.0 (1767.77)
  Week 33 to 34: number analyzed (Participants) | 1 | 3
  Week 33 to 34 | 12000.0 (NA) — Only 1 participant analyzed at this time point. | 2816.7 (1877.72)
  Week 35 to 36: number analyzed (Participants) | 1 | 0
  Week 35 to 36 | 12000.0 (NA) — Only 1 participant analyzed at this time point. |
  Week 37 to 38: number analyzed (Participants) | 2 | 2
  Week 37 to 38 | 4795.0 (4532.55) | 3500.0 (2828.43)
  Week 39 to 40: number analyzed (Participants) | 2 | 2
  Week 39 to 40 | 26795.0 (35645.25) | 2375.0 (883.88)
  Week 41 to 42: number analyzed (Participants) | 1 | 1
  Week 41 to 42 | 24000.0 (NA) — Only 1 participant analyzed at this time point. | 1500.0 (NA) — Only 1 participant analyzed at this time point.
  Week 43 to 44: number analyzed (Participants) | 1 | 1
  Week 43 to 44 | 20000.0 (NA) — Only 1 participant analyzed at this time point. | 1750.0 (NA) — Only 1 participant analyzed at this time point.
  Week 45 to 46: number analyzed (Participants) | 1 | 1
  Week 45 to 46 | 20000.0 (NA) — Only 1 participant analyzed at this time point. | 5000.0 (NA) — Only 1 participant analyzed at this time point.
  Week 47 to 48: number analyzed (Participants) | 1 | 1
  Week 47 to 48 | 20000.0 (NA) — Only 1 participant analyzed at this time point. | 7500.0 (NA) — Only 1 participant analyzed at this time point.
  Week 49 to 50: number analyzed (Participants) | 1 | 0
  Week 49 to 50 | 24000.0 (NA) — Only 1 participant analyzed at this time point. |
  Week 51 to 52: number analyzed (Participants) | 1 | 0
  Week 51 to 52 | 20000.0 (NA) — Only 1 participant analyzed at this time point. |

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 52 weeks after dosing (Cohort 1) or 44 weeks after dosing (Cohort 2).
Description: TEAEs are presented. A TEAE was defined as any event not present before exposure to study product or any event already present that worsened in severity or increased in frequency after exposure to study product. Due to concerns related to participant re-identification in this study, events are presented by system organ class only.
Arm/Group | DTX101, Cohort 1 | DTX101, Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DTX101, Cohort 1 (N=3) | DTX101, Cohort 2 (N=3)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DTX101, Cohort 1 (N=3) | DTX101, Cohort 2 (N=3)
Investigations (Investigations) | 1 | 3
Infections and infestations (Infections and infestations) | 1 | 2
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 | 1
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 | 1
Gastrointestinal disorders (Gastrointestinal disorders) | 1 | 1
General disorders and administration site conditions (General disorders) | 1 | 1
Nervous system disorders (Nervous system disorders) | 1 | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Eye disorders (Eye disorders) | 0 | 1
Psychiatric disorders (Psychiatric disorders) | 0 | 1
Vascular disorders (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
After review of the DTX101 Phase 1/2 clinical trial data, a decision was made to discontinue the development of DTX101. The discontinuation was not due to any safety concerns related to DTX101.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2015-09-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT02618915/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT02618915/SAP_001.pdf